CLINICAL TRIAL: NCT03465072
Title: Abnormal Vascular, Metabolic, and Neural Function During Exercise in Heart Failure With Preserved Ejection Fraction
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The first major aim of this project has been accomplished. Currently, this project is temporarily on hold while other projects are prioritized.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin Levine, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU 082017-038
Record Dates: First submitted 2018-02-20; First posted 2018-03-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Normal Ejection Fraction
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise training (Experimental): 8 Weeks exercise training 3x per week 30-40 minutes per session
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — 8 weeks, 3 times per week, 30-40 minutes

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) accounts for approximately half of the heart failure population in the United States. The primary chronic symptom in patients with HFpEF is severe exercise intolerance quantified as reduced peak oxygen uptake during whole body exercise (peak V̇O2). To date, studies have focused almost exclusively on central cardiac limitations of peak V̇O2 in HFpEF. However, in stark contrast to heart failure with reduced ejection fraction (HFrEF), drug therapies targeting central limitations have invariably failed to improve peak V̇O2, quality of life, or survival in HFpEF. Emerging evidence from our lab suggests reduced skeletal muscle oxidative capacity may contribute to exercise intolerance in HFpEF patients. However, the mechanisms responsible for peripheral metabolic inefficiency remain unclear. Reduced blood flow (oxygen delivery), and slowed oxygen uptake kinetics (O2 utilization) may both contribute to reduced peripheral oxidative capacity. Importantly, reduced oxidative capacity may result in increased production of metabolites known to activate muscle afferent nerves and stimulate reflex increases in muscle sympathetic (vasoconstrictor) nervous system activity (MSNA). However, to date there have been no studies specifically investigating the contribution of peripheral metabolic and neural impairments to reduced exercise capacity in HFpEF. The overall aim of this proposal will be 1) to identify impairments in peripheral vascular, metabolic, and sympathetic neural function and 2) to assess the ability of small muscle mass (knee extensor, KE) training, specifically targeting these peripheral skeletal muscle deficiencies, to improve aerobic capacity and exercise tolerance in HFpEF.

GLOBAL HYPOTHESIS 1: HFpEF patients will demonstrate reduced skeletal muscle oxygen delivery, slowed oxygen uptake kinetics, and elevated resting and metaboreflex mediated MSNA.

Hypothesis 1.1: The vasodilatory response to knee extensor exercise will be impaired in HFpEF patients.

Specific Aim 1.1: To measure the immediate rapid onset vasodilatory response to muscle contraction, as well as the dynamic onset, and steady state vasodilatory responses to dynamic KE exercise.

Hypothesis 1.2: Skeletal muscle oxygen uptake kinetics will be slowed in HFpEF.

Specific Aim 1.2: To measure pulmonary oxygen uptake kinetics during isolated KE exercise in order to isolate peripheral impairments in metabolic function independent of any central impairment.

Hypothesis 1.3: HFpEF patients will demonstrate elevated MSNA at rest, and exaggerated metaboreflex sensitivity during exercise.

Specific Aim 1.3: To test this hypothesis the investigators will measure MSNA from the peroneal nerve at rest, and during post exercise ischemia to directly assess metaboreflex sensitivity in HFpEF.

GLOBAL HYPOTHESIS 2: Isolating peripheral adaptations to exercise training using single KE exercise training will improve peripheral vascular, metabolic, and neural function and result in greater functional capacity in HFpEF.

Hypothesis 2.1: Isolated KE exercise training will improve the vasodilatory response to exercise, speed oxygen uptake kinetics, and reduce MSNA at rest HFpEF.

Specific Aim 2.1: The assessments of vascular, metabolic, and neural function proposed in hypothesis 1 will be repeated after completing 8 weeks of single KE exercise training.

Hypothesis 2.2: Single KE exercise training will improve whole body exercise tolerance, peak V̇O2, and functional capacity in HFpEF.

Specific Aim 2.2: To test this hypothesis the investigators will measure maximal single KE work rate, V̇O2 kinetics and peak V̇O2 during cycle exercise, as well as distance covered in the six minute walk test.

DETAILED DESCRIPTION:
Protocol 1.1: To test hypothesis 1.1 the investigators will measure rapid onset vasodilation in response to a single KE contraction as a marker of vascular responsiveness to muscle contraction, as well as the dynamic onset, and steady state vasodilatory responses to continuous KE exercise. The rapid onset vasodilatory (ROV) response to a brief (1-second) single isometric knee extension contraction will be measured as described by our collaborators50. Subjects will perform single contractions at 5, 10 or 20% of their maximal voluntary contraction (MVC). Beat-by-beat local vascular responses (i.e. femoral blood flow; FBF and vascular conductance; FVC) will be recorded continuously for 30-seconds with the initial response (first un-interrupted cardiac cycle post-contraction), peak response (maximal increase), latency (time to peak response) and area under the curve (total vasodilator response across 30-seconds) analyzed to fully characterize ROV in HFpEF. Additionally, the vascular and hemodynamic response to dynamic KE exercise (beat-by-beat onset and steady state FBF and FVC) will be measured from the onset of exercise for six minutes at submaximal work rates (10, 15 W, and 60% maximal work rate). These trials will be performed individually and with 20 minutes of rest between conditions to ensure that patients will be able to complete each of these trials. In addition to local vascular hemodynamics, systemic hemodynamics (HR, MAP, CO, SV) will be monitored throughout to confirm that any alterations in local blood flow are independent of central cardiovascular adjustments (See Fig. 2, Day 2)

Hypothesis 1.2: Skeletal muscle V̇O2 kinetics will be slowed in HFpEF.

Protocol 1.2: Breath-by-breath pulmonary V̇O2 kinetics will be measured during cycle exercise at a relatively light work rate of 20 W (~30% V̇O2 peak) to characterize V̇O2 kinetics where there is no cardiac limitation, allowing for a submaximal assessment of "peripheral" oxidative efficiency during large muscle mass exercise. During cycle exercise, V̇O2 kinetics will be measured in conjunction near infrared spectroscopy as a marker of the coupling between oxygen delivery and demand (see Fig. 2, Day 3).

Hypothesis 1.3: HFpEF patients will demonstrate elevated MSNA at rest, and exaggerated metaboreflex sensitivity during exercise.

Protocol 1.3: Microneurography will be used to measure multi-unit muscle sympathetic nerve discharge in subjects at rest, during dynamic knee extension exercise (30, 40% MVC), and during 2 minutes and 15 seconds of post-exercise ischemia (PEI) achieved via inflation of a blood pressure cuff to supra-systolic pressure. This approach allows for experimental isolation of the metaboreflex contribution to changes in MSNA and hemodynamics by preventing washout of metabolites produced by muscle contraction during exercise. Importantly, the sympathetic response is independent of the confounding activation of the mechanoreflex or central command as muscle contractions are no longer being performed. A cold pressor test will be utilized to confirm specific sensitivity to the metaboreflex and not generalized sensitivity to sympathoexcitatory stimuli. Multi-unit post-ganglionic MSNA will be recorded from the peroneal nerve using standard microneurographic techniques and quantified as burst frequency (bursts/min), burst incidence (burst/100 cardiac cycles) and total activity (burst frequency x mean burst amplitude).

Experimental Series 2 - Global Hypothesis 2: isolating peripheral adaptations to exercise training using single KE exercise training will improve peripheral vascular, metabolic, and neural function and result in greater functional capacity in HFpEF.

Approach: Hypothesis 2.1: Isolated KE exercise training will improve the vasodilatory response to exercise, speed V̇O2 kinetics, and reduce MSNA at rest HFpEF.

Protocol 2.1: 1) Vascular response: ROV will be assessed as described in protocol 1. Subjects will perform single contractions at 5, 10 or 20% of their pre- and post-testing maximal voluntary contraction (MVC). The peripheral hemodynamic response to dynamic KE exercise (beat-by-beat onset and steady state) will be measured continuously from the onset of exercise for six minutes at the same absolute (10, and 15 W) and relative (60% of post-intervention maximal work rate) exercise intensities. Local vascular (FBF, FVC) and systemic (HR, MAP, CO, SV) hemodynamics will be monitored throughout these trials to confirm that any alterations in local blood flow are independent of central cardiovascular adaptations (See Fig 2, Day 2). 2) V̇O2 Kinetics: Breath-by-breath Pulmonary V̇O2 kinetics will be measured during isolated single KE exercise and during upright cycle exercise. Dynamic KE exercise will be performed for six minutes at the same absolute submaximal work rates (10 and 15 W) as well as the same relative (60% post-intervention maximal work rate; see Fig 2, Day 2) in conjunction with beat-by-beat blood flow measures. Additionally, V̇O2 kinetics will be assessed during mild intensity cycle exercise at 20 W and utilized as a marker of intervention efficacy as discussed above (see Fig. 2, Day 3). 3) MSNA: Microneurography will be used to measure multi-unit muscle sympathetic nerve discharge in subjects at rest, during knee extension exercise, and PEI (See Fig 2, Day 3).

Hypothesis 2.2: Single KE exercise training will improve whole body exercise tolerance, peak V̇O2, and functional capacity in HFpEF.

Protocol 2.2: In addition to submaximal V̇O2 kinetics: maximal KE work rate, peak V̇O2 during cycle exercise, and performance in the 6-minute walk test will be re-evaluated after isolated quadriceps exercise training in the same manner as prior to the intervention (see specific exercise training protocol below).

ELIGIBILITY:
All subjects will be >65 years of age. The controls will be screened carefully for hypertension and cardiac disease, including structural heart and hemodynamically significant obstructive coronary disease, using a history, physical examination, and resting and post-exercise transthoracic echocardiograms. Additional exclusion criteria for this group will include valvular heart disease, atrial flutter/ fibrillation, renal insufficiency, chronic lung disease, regular cigarette smoking within the past 10 years, and cardiovascular medication. Subjects demonstrating greater than moderate levels of activity > 2 days per week will not be allowed to participate, as chronic high levels of physical activity could potentially impact the primary outcome variables.

* HFpEF Inclusion Criteria:
* Patients will be > 65 years old
* We will use a modification of the European Guidelines for the diagnosis of HFpEF to select the patient population.
* The key components of these guidelines include:

  * signs and symptoms of heart failure;
  * b) an ejection fraction > 0.50; and
  * c) objective evidence of diastolic dysfunction. To satisfy the first criteria, we will use the Framingham criteria (dyspnea, orthopnea, PND, edema); however we will require objective evidence of congestion including
* chest X-ray,
* elevated BNP,
* or elevated PCWP (pulmonary capillary wedge pressure) or
* LVEDP (left ventricular end-diastolic pressure) > 16 mmHg; for the second, we will accept echo, nuclear or catheter documentation; and for
* we will require a depressed tissue Doppler mitral annular velocity < 7.5 cm/s along with PCWP > 16 mmHg if available.

HFpEF Exclusion Criteria:

* underlying valvular or congenital heart disease;
* restrictive or infiltrative cardiomyopathy;
* acute myocarditis;
* NYHA Class IV CHF, or CHF that cannot be stabilized on medical therapy;
* other condition that would limit the patient's ability to complete the protocol;
* manifest ischemic heart disease.
* Patients with CABG or previous history of atrial fibrillation will be allowed to participate, though for safety reasons, patients on Coumadin will be excluded.
* All patients must be in sinus rhythm without a left bundle branch block at the time of study, and be off beta blockers or non-dihydropyridine Ca++ blockers for at least 5 half-lives. β blockers will be weaned over 3-5 days and additional doses of vasodilators added to control blood pressure if necessary. Drugs that affect the renin-angiotensin-aldosterone system and diuretics will be maintained.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Muscle sympathetic nervous system activity | Change in muscle sympathetic nervous system activity after 8 weeks of exercise training
  Sympathetic neural activity measured during exercise
VO2 onset kinetics | Change in VO2 onset kinetics after 8 weeks of exercise training
  Rise in oxygen uptake during exercise

SECONDARY OUTCOMES:
Reactive hyperemia | Change in Reactive hyperemia after 8 weeks of exercise training
  Blood flow in response to ischemia
Exercise hyperemia | Change in exercise hyperemia after 8 weeks of exercise training
  Blood flow response to exercise

CONTACTS AND LOCATIONS:
Locations (1):
- The Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No